CLINICAL TRIAL: NCT01139229
Title: Phase III Study of Hybrid-everted Versus Hand-sewn of Stapled Esophagogastrostomy in Prevention of Anastomotic Stricture
Brief Title: Hybrid-everted Versus Hand-sewn or Stapled Esophagogastrostomy in Prevention of Anastomotic Stricture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Long-Qi Chen, Professor, Department of Thoracic and Cardiovascular Surgery, West China Hospital of Sichuan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCH20070901
Record Dates: First submitted 2010-06-03; First posted 2010-06-08 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Esophageal Neoplasms; Surgical Stomas
Keywords: Esophagogastrostomy; Circular everted anastomosis; Side-side anastomosis; Randomized clinical trial
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HE group (Other)
  Interventions: Other: hybrid everted esophagogastric anastomosis
- HS group (Other)
  Interventions: Other: the conventional hand-sewn anastomosis
- SA group (Other)
  Interventions: Other: a stapled anastomosis

INTERVENTIONS:
Other: hybrid everted esophagogastric anastomosis
  Other Names: no other names
  Arms: HE group
Other: the conventional hand-sewn anastomosis
  Other Names: no other names
  Arms: HS group
Other: a stapled anastomosis
  Other Names: no other names
  Arms: SA group

SUMMARY:
The investigators improved the hybrid everted esophagogastrostomy and expected to prevent the incidence of anastomotic stricture. The purpose of this study is to determine the clinical value of this kind of operation type, and analyzes the clinicopathological factors causing the postoperative complications.

DETAILED DESCRIPTION:
This randomized clinical trial compared a hybrid everted esophagogastric anastomosis with conventional hand-sewn or stapled esophagogastrostomy for prevention of anastomotic stricture. The patients were completely randomized to receive either a hybrid everted esophagogastric anastomosis (HE group), or the conventional hand-sewn (HS group), or a stapled (SA group) anastomosis, after the removal of esophageal tumor. The primary outcome measured the incidence of anastomotic stricture at 3 months after the operation (defined as the diameter of the anastomotic orifice <= 0.8 cm on esophagogram), analyzed by intention-to-treat.

ELIGIBILITY:
Inclusion Criteria:

* pathologically diagnosed esophageal neoplasms
* undergoing the Esophagogastrostomy

Exclusion Criteria:

* the patients with previous the upper gastrointestinal tract surgery
* the esophageal carcinoma patients with previous neoadjuvant chemotherapy
* the esophageal carcinoma complicated other esophagogastric diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2007-11; Primary Completion 2007-11 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
the incidence of anastomotic stricture | three months
  the anastomotic stricture is defined as the diameter of the anastomotic orifice <= 0.8 cm on esophagogram

SECONDARY OUTCOMES:
The grades of dysphagia | three months
  0:No dysphagia on solid diet
  1. dysphagia on solid diet
  2. dyspahgia on semi-solid diet
  3. dysphagia on fluid diet
  4. dysphagia with water swallowing
the grades of acid regurgitation | three months
  0:no reflux on semi-supine position
  1. postprandial reflux on semi-supine position
  2. reflux with empty stomatch on semi-supine position
  3. postprandial reflux on upright position
  4. reflux with empty stomach on upright positino
the clinicopathological parameters in relation to postoperative complications | three months

CONTACTS AND LOCATIONS:
Overall Officials: Qi L Chen, Study Chair — the Department of Cardiothoracic Surgery, Huaxi Hospital of Sichuan University

REFERENCES:
- [Result] Law S, Fok M, Chu KM, Wong J. Comparison of hand-sewn and stapled esophagogastric anastomosis after esophageal resection for cancer: a prospective randomized controlled trial. Ann Surg. 1997 Aug;226(2):169-73. doi: 10.1097/00000658-199708000-00008. PMID 9296510
- [Result] Behzadi A, Nichols FC, Cassivi SD, Deschamps C, Allen MS, Pairolero PC. Esophagogastrectomy: the influence of stapled versus hand-sewn anastomosis on outcome. J Gastrointest Surg. 2005 Nov;9(8):1031-40; discussion 1040-2. doi: 10.1016/j.gassur.2005.06.025. PMID 16269373
- [Result] Moher D, Schulz KF, Altman D; CONSORT Group. The CONSORT Statement: revised recommendations for improving the quality of reports of parallel-group randomized trials 2001. Explore (NY). 2005 Jan;1(1):40-5. doi: 10.1016/j.explore.2004.11.001. PMID 16791967
- [Result] Zhu ZJ, Zhao YF, Chen LQ, Hu Y, Liu LX, Wang Y, Kou YL. Clinical application of layered anastomosis during esophagogastrostomy. World J Surg. 2008 Apr;32(4):583-8. doi: 10.1007/s00268-007-9396-5. PMID 18210181
- [Result] Laterza E, de' Manzoni G, Veraldi GF, Guglielmi A, Tedesco P, Cordiano C. Manual compared with mechanical cervical oesophagogastric anastomosis: a randomised trial. Eur J Surg. 1999 Nov;165(11):1051-4. doi: 10.1080/110241599750007883. PMID 10595609
- [Derived] Wang WP, Gao Q, Wang KN, Shi H, Chen LQ. A prospective randomized controlled trial of semi-mechanical versus hand-sewn or circular stapled esophagogastrostomy for prevention of anastomotic stricture. World J Surg. 2013 May;37(5):1043-50. doi: 10.1007/s00268-013-1932-x. PMID 23381675